CLINICAL TRIAL: NCT03429816
Title: Molecular Outcome Prediction of Neoadjuvant Systemic Treatment in Esophagogastric Carcinoma
Brief Title: OPPOSITE: Outcome Prediction of Systemic Treatment in Esophagogastric Carcinoma
Acronym: OPPOSITE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Heidelberg (Other)
Collaborators: University Hospital Dresden (Other); German Cancer Research Center (Other)
Responsible Party: Principal Investigator, Georg Martin Haag, NCT, Dep. Medical Oncology, University Hospital Heidelberg
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: OPPOSITE
Record Dates: First submitted 2018-02-05; First posted 2018-02-12 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Gastric Neoplasm; Gastroesophageal Junction Adenocarcinoma; Esophageal Adenocarcinoma; Gastric Adenocarcinoma; Esophageal Neoplasms
MeSH Terms: conditions — Stomach Neoplasms; Adenocarcinoma Of Esophagus; Esophageal Neoplasms | interventions — Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Interventional Arm (Experimental): Patients with locally advanced, resectable gastric or esophagogastric junction adenocarcinoma will receive a biopsy of the primary tumor, followed by standard-of care neoadjuvant systemic treatment; after neoadjuvant therapy tumor biopsies will be taken from different sites of the resection specimen.
  Organoid cultures of pre-treatment tumor biopsies will be established and exposed to the same chemotherapy as the corresponding patient; in vitro response to treatment will be correlated with the in vivo response of patients.
  Whole genome, methylome and RNA sequencing of tumors biopsies and organoids will be performed prior to as well as after systemic treatment.
  Interventions: Procedure: Biopsy

INTERVENTIONS:
Procedure: Biopsy — Patients with locally advanced, resectable gastric or esophagogastric junction adenocarcinoma will receive a biopsy of the primary tumor, followed by standard-of care neoadjuvant systemic treatment; after neoadjuvant therapy tumor biopsies will be taken from different sites of the resection specimen.

SUMMARY:
Patients with locally advanced, resectable gastric or esophagogastric junction adenocarcinoma will receive a biopsy of the primary tumor, followed by standard-of care neoadjuvant systemic treatment; after neoadjuvant therapy tumor biopsies will be taken from different sites of the resection specimen.

* Aim 1: Organoid cultures of pre-treatment tumor biopsies will be established and exposed to the same chemotherapy as the corresponding patient; in vitro response to treatment will be correlated with the in vivo response of patients.
* Aim 2: Whole genome, methylome and RNA sequencing of tumors biopsies and organoids will be performed prior to as well as after systemic treatment. Histological and clinical outcome will be correlated with molecular subtypes.

ELIGIBILITY:
Inclusion Criteria:

Histologically confirmed, resectable adenocarcinoma of the GEJ (type I-III) or the stomach (cT2, cT3,cT4, any cN category, M0), or any cT cN+ M0 with the following specifications:

* ECOG-Score ≤ 2
* Patient is fit to undergo surgery (either subtotal or total gastrectomy, transhiatal or abdominothoracic esophagectomy)
* No preceding cytotoxic or targeted therapy
* No prior partial or complete tumor resection
* Exclusion of distant metastasis by CT or MRI of thorax and abdomen, and optionally bone scan (if osseous lesions are suspected due to clinical signs)

Exclusion Criteria:

* Patients with distant metastasis
* Known hypersensitivity against components of the neoadjuvant systemic treatment
* Documented history of congestive heart failure NYHA ≥III, myocardial infarction within the past 3 months before the start of neoadjuvant treatment
* Uncontrollable high-risk cardiac arrhythmia, e.g. significant ventricular arrhythmia
* Past or current history of other malignancies not curatively treated and without evidence of disease for more than 5 years, except for curatively treated early stage cancers such as basal cell carcinoma of the skin and in situ carcinoma of the cervix or the bladder.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2018-04-15 (Actual); Primary Completion 2021-11-01 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
Aim 1: Correlation of in-vitro response in the organoid model with histological regression in the resected tumor | 1 year
  Correlation of in-vitro response to cytotoxic chemotherapy in the patient-derived organoid model with histological regression in the resected specimen and analysis of reliability of this organoid model in predicting patients' response to neoadjuvant chemotherapy.
Aim 2: Correlation of molecular subtypes with histological response after neoadjuvant therapy in patients | 1 year
  Prognostic impact of the molecular subtypes on histological response to neoadjuvant chemotherapy in patients will be modeled using the logistic regression.

SECONDARY OUTCOMES:
Aim 1: Correlation of in-vitro response in the organoid model with relapse-free survival | maximum 5 years
  The possible prognostic impact of in-vitro response in the organoid model on relapse-free survival will be investigated using the Cox proportional hazards models.
Aim 2: Correlation of molecular subtypes with relapse-free survival | maximum 5 years
  The possible prognostic impact of molecular subtypes on relapse-free survival will be investigated using the Cox proportional hazards models.

OTHER OUTCOMES:
Aim 1: Correlation of in-vitro response in the organoid model with overall survival | maximum 5 years
  The possible prognostic impact of in-vitro response in the organoid model on overall survival will be investigated using the Cox proportional hazards models.
Aim 2: Correlation of molecular subtypes with overall survival | maximum 5 years
  The possible prognostic impact of molecular subtypes on overall survival will be investigated using the Cox proportional hazards models.

CONTACTS AND LOCATIONS:
Overall Officials: Georg Martin Haag, Principal Investigator — NCT, University Hospital Heidelberg
Locations (2):
- Germany (2):
  - University Hospital Dresden, Dresden
  - National Center for Tumor Diseases, University Hospital Heidelberg, Heidelberg